CLINICAL TRIAL: NCT02064972
Title: Evaluation of Circulating Endothelial Cells (CEC) as a Marker of Endothelial Damage in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT): Correlation With the Occurrence of Graft-versus-Host Disease (GvHD)
Brief Title: CEC Count Changes to Support GvHD Diagnosis.
Acronym: ALLOCEC
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Janssen Diagnostics, LLC (Industry)
Responsible Party: Principal Investigator, Camillo Almici MD, M.D., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP 1574
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Graft vs Host Disease; Complications of Organ Transplant Stem Cells; Endothelial Dysfunction
Keywords: Graft vs Host Disease; Hematopoietic Stem Cell Transplant; Biological Marker; Circulating Endothelial Cells; Endothelial Dysfunction
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing allo-HSCT, who manifest GvHD.: Patients undergoing allo-HSCT, that manifest GvHD. Patients undergoing allo-HSCT will have CEC count performed at the following timepoints: T1 (baseline), T2 (pre-transplant), T3 (engraftment), T4 (GvHD onset) and T5 (post-GvHD). All patients will also be checked for CEC at day + 28.
  Interventions: Other: Patients undergoing allo-HSCT, who manifest GvHD.

INTERVENTIONS:
Other: Patients undergoing allo-HSCT, who manifest GvHD. — Changes in CEC counts in relation to GvHD ONSET

SUMMARY:
In consideration of the fact that the vascular endothelium has been shown to be a target of GvHD in early stage and that the count of CEC may represent a marker of endothelial damage, we want to evaluate the changes in CEC counts of patients affected by hematological disorders undergoing allo-HSCT, as a function of endothelial damage. We will enroll 50 patients affected by hematologic disorders undergoing allo-HSCT. Peripheral blood will be drawn before (T1, baseline) and at the end of the conditioning regimen (T2, pre-transplant), upon confirmation of hematopoietic recovery (T3, engraftment) and thereafter at onset of GVHD (GVHD T4) and one week after the start of steroid therapy (T5, post-GvHD). All patients will also be checked for CEC at day + 28. CEC enumeration will be performed by using the CellSearch® System and a flowcytometry procedure.

Through the conduct of this study, we expect to confirm our preliminary results on a larger series of patients, and to evaluate the predictive role of CEC on the occurrence of GvHD and prognostic response to treatment of GvHD. The possibility of early identification of patients who do not respond to traditional treatments of GvHD, and for this reason at a higher risk of morbidity and mortality, may allow greater individualization of the therapeutic program, for example with the introduction as early as possible of alternative treatments. In addition, the identification of patients at higher risk of non-responsiveness to steroid treatment, would allow, through a closer monitoring, the early introduction of additional treatment before the development of resistance/refractoriness to treatment of GvHD.

The present study takes the form of a prospective study. The primary endpoint is the identification and enumeration of CECs in peripheral blood of patients with hematological disorder undergoing allo-HSCT, as a function of endothelial damage. The secondary endpoint is to define the prognostic and predictive value of the changes of CEC counts on the diagnosis of GvHD and response to treatment.

DETAILED DESCRIPTION:
The endothelial damage is a characteristic common to several complications of vascular origin that may occur in the course of allo-HSCT (GVHD, IPS, VOD, TMA). The diagnosis of vascular complications represents an interesting challenge, but unfortunately limited by the fact that the markers of endothelial damage are extremely scarce. In particular, the plasmatic dosage of von Willebrand factor, thrombomodulin and adhesion molecules generated results difficult to use for a potential application for routine diagnostics for the high degree of non-specificity and the potential influence on the assay by co-morbid conditions related to the recipient. Much more promising methods appear to be those that are based on the evaluation of microparticles derived from endothelial cells (EMP) or the direct counting of circulating endothelial cells (CEC). Recently, the EMP were assessed by flow cytometry (annexin V-FITC and anti-CD62-PE) in 19 patients undergoing allo-HSCT, showing an increase in patients with acute GvHD grade ≥ I, compared to patients that did not display GvHD. In addition, the evaluation of EMP did not appear to be affected by the radio-chemotherapy conditioning regimen. This method is, however, burdened with a procedural complexity and a certain degree of non-specificity due to the fact that the microparticles can be released by endothelial cells as well as also from platelets, red blood cells and leukocytes.

Currently, the direct counting of the CEC seems to be the most reliable ways to assess the degree of endothelial damage. The finding of elevated numbers of CEC has been shown to reflect the extent of endothelial damage in numerous pathologies of autoimmune nature, but are still preliminary data in the course of allo-HSCT. Woywodt et al. demonstrated in patients with ANCA-positive vasculitis a correlation between the number of CEC and the degree of disease activity and response to treatment. Moreover, the number of CEC correlates, in patients undergoing renal transplantation, with the risk of organ rejection. In the course of allo-HSCT, the same authors have shown a correlation between the number of CEC and endothelial damage induced by radio-chemotherapy conditioning regimen. However, the lack of a standardized method, the use of manual procedures of immunoselection, the lack of consensus on the identification of CEC represent limiting factors for routine application.

The present study takes the form of a prospective study. The primary endpoint is the identification and enumeration of CECs in peripheral blood of patients with hematological disorders undergoing allo-HSCT, as a function of endothelial damage. The secondary endpoint is to define the prognostic and predictive value of CEC counts changes on the diagnosis of GvHD and on the response to treatment.

Peripheral blood (PB) will be drawn before (T1, baseline) and at the end of the conditioning regimen (T2, pre-transplant), upon confirmation of hematopoietic recovery (T3, engraftment) and thereafter at onset of GVHD (GVHD T4) and one week after the start of steroid therapy (T5, post-GvHD) for the control of GvHD. All patients will also be checked for CEC at day + 28.

The peripheral blood for counting CEC will be collected, respectively, in the CellSave Preservative Tube (Veridex, J & J, USA), containing a preservative for the stabilization of the cells at room temperature, for counting with the CellSearch® System and in CBC tube containing K2EDTA, for counting by flow cytometry.

By the CellSearch® System an event will be classified as CEC when its morphology is consistent with that of a cell and simultaneously shows the following phenotype: CD146+, CD105+, DAPI+ and CD45-. By the flowcytometry procedure, after staining of cells with lyophilized antibodies of the Endo Panel tube (CD146, 7-AAD, CD34, CD309, CD45) 4x106 events in the lympho-monocyte gate will be immediately aquired at flowcytometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological disorders undergoing allo-HSCT,
* Age 18-65 years.
* Sign of written informed consent form at the time of study entry.

Exclusion Criteria:

* No candidates to allo-HSCT.
* Patients under the age of 18 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, affected by hematologic disorders, undergoing allo-HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline (Timepoint 1) in Circulating Endothelial Cell (CEC) count at GvHD onset (Timepoint 4) | Basal (Timepoint 1) versus GvHD onset (Timepoint 4)
  CEC count changes will be evaluated between baseline and time of GvHD onset, within day + 100 post-transplant. In our preliminary series of 40 patients GvHD have manifested at a median of 27 days post-transplant (range 15-103).

SECONDARY OUTCOMES:
Changes from baseline (Timepoint 1) in Circulating Endothelial Cell (CEC) count at time of transplant (Timepoint 2) | Basal (Timepoint 1) versus pre-transplant (Timepoint 2)
  CEC count changes will be evaluated between baseline and pre-transplant, which usually is in the range of 5-8 days.
Changes from baseline (Timepoint 1) in Circulating Endothelial Cell (CEC) count at time of engraftment (Timepoint 3). | Basal (Timepoint 1) versus engraftment (Timepoint 3)
  CEC count changes will be evaluated between baseline and time of engraftment. In our preliminary series of 40 patients engraftment occurred at a median of 22 days post-transplant (range 14-31).
Changes from GvHD onset (Timepoint 3) in Circulating Endothelial Cell (CEC) count at one week after the start of steroid therapy (Timepoint 5). | GvHD onset (Timepoint 3) versus one week after the start of steroid therapy (Timepoint 5)
  CEC count changes will be evaluated between GVHD onset and one week after steroid therapy

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Almici, M.D., Principal Investigator — Transfusion Medicine, Spedali Civili Brescia, Italy
Locations (1):
- A.O. Spedali Civili of Brecia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analysed during the current study will be available from the corresponding author on reasonable request after the publication of results.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of results
Access Criteria: Request to Principal Investigator

REFERENCES:
- [Background] Rowand JL, Martin G, Doyle GV, Miller MC, Pierce MS, Connelly MC, Rao C, Terstappen LW. Endothelial cells in peripheral blood of healthy subjects and patients with metastatic carcinomas. Cytometry A. 2007 Feb;71(2):105-13. doi: 10.1002/cyto.a.20364. PMID 17226859
- [Background] Woywodt A, Scheer J, Hambach L, Buchholz S, Ganser A, Haller H, Hertenstein B, Haubitz M. Circulating endothelial cells as a marker of endothelial damage in allogeneic hematopoietic stem cell transplantation. Blood. 2004 May 1;103(9):3603-5. doi: 10.1182/blood-2003-10-3479. Epub 2004 Jan 8. PMID 14715625
- [Background] Damani S, Bacconi A, Libiger O, Chourasia AH, Serry R, Gollapudi R, Goldberg R, Rapeport K, Haaser S, Topol S, Knowlton S, Bethel K, Kuhn P, Wood M, Carragher B, Schork NJ, Jiang J, Rao C, Connelly M, Fowler VM, Topol EJ. Characterization of circulating endothelial cells in acute myocardial infarction. Sci Transl Med. 2012 Mar 21;4(126):126ra33. doi: 10.1126/scitranslmed.3003451. PMID 22440735
- [Background] Chen YB, Cutler CS. Biomarkers for acute GVHD: can we predict the unpredictable? Bone Marrow Transplant. 2013 Jun;48(6):755-60. doi: 10.1038/bmt.2012.143. Epub 2012 Aug 6. PMID 22863728
- [Background] Carreras E, Diaz-Ricart M. The role of the endothelium in the short-term complications of hematopoietic SCT. Bone Marrow Transplant. 2011 Dec;46(12):1495-502. doi: 10.1038/bmt.2011.65. Epub 2011 Apr 4. PMID 21460864
- [Background] Penack O, Socie G, van den Brink MR. The importance of neovascularization and its inhibition for allogeneic hematopoietic stem cell transplantation. Blood. 2011 Apr 21;117(16):4181-9. doi: 10.1182/blood-2010-10-312934. Epub 2011 Jan 21. PMID 21258010
- [Background] Almici C, Skert C, Verardi R, Di Palma A, Bianchetti A, Neva A, Braga S, Malagola M, Turra A, Marini M, Russo D. Changes in circulating endothelial cells count could become a valuable tool in the diagnostic definition of acute graft-versus-host disease. Transplantation. 2014 Oct 15;98(7):706-12. doi: 10.1097/TP.0000000000000385. PMID 25119132
- [Background] Lanuti P, Rotta G, Almici C, Avvisati G, Budillon A, Doretto P, Malara N, Marini M, Neva A, Simeone P, Di Gennaro E, Leone A, Falda A, Tozzoli R, Gregorj C, Di Cerbo M, Trunzo V, Mollace V, Marchisio M, Miscia S. Endothelial progenitor cells, defined by the simultaneous surface expression of VEGFR2 and CD133, are not detectable in healthy peripheral and cord blood. Cytometry A. 2016 Mar;89(3):259-70. doi: 10.1002/cyto.a.22730. Epub 2015 Aug 25. PMID 26305912
- [Derived] Almici C, Neva A, Skert C, Bruno B, Verardi R, Di Palma A, Bianchetti A, Braga S, Piovani G, Cancelli V, Omede P, Baeten K, Rotta G, Russo D, Marini M. Counting circulating endothelial cells in allo-HSCT: an ad hoc designed polychromatic flowcytometry-based panel versus the CellSearch System. Sci Rep. 2019 Jan 14;9(1):87. doi: 10.1038/s41598-018-36442-9. PMID 30643152
- [Derived] Almici C, Skert C, Bruno B, Bianchetti A, Verardi R, Di Palma A, Neva A, Braga S, Piccinelli G, Piovani G, Malagola M, Bernardi S, Giaccone L, Brunello L, Festuccia M, Baeten K, Russo D, Marini M. Circulating endothelial cell count: a reliable marker of endothelial damage in patients undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2017 Dec;52(12):1637-1642. doi: 10.1038/bmt.2017.194. Epub 2017 Sep 11. PMID 28892085